CLINICAL TRIAL: NCT05174780
Title: Clinical Evaluation of A Innovative Spectacle Lens in Slowing Myopia Progression
Brief Title: Myopia Control With a Innovative Spectacle Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WS10246
Record Dates: First submitted 2021-12-13; First posted 2022-01-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Myopia
Keywords: spectacle; myopia control; myopia; HAL; Stellest; Essilor
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Innovative myopia control spectacle lens (Experimental)
  Interventions: Device: innovative myopia control spectacle lens
- Single vision spectacle lens (Placebo Comparator)
  Interventions: Device: Single vision spectacle lens

INTERVENTIONS:
Device: innovative myopia control spectacle lens — using a innovative spectacle lens to control myopia progression
  Arms: Innovative myopia control spectacle lens
Device: Single vision spectacle lens — single vision spectacle lens for myopia and astigmatism correction
  Arms: Single vision spectacle lens

SUMMARY:
The purpose of this study is to demonstrate that the test spectacle lens is safe and effective in slowing myopia progression in children.

ELIGIBILITY:
Inclusion Criteria:

* Equal to or greater than 6 years and not older than 12 years at time of informed consent and assent.
* Spherical equivalent refractive error (SER) by manifest refraction between -0.75 and -4.50 D in each eye.
* Astigmatism, if present, of not more than 1.50 D.
* Difference in SER between the two eyes (Anisometropia) by manifest refraction not more than 1.00 D.
* Best corrected visual acuity in each eye equal to or better than +0.10 logMAR (≥ 20/25 as Snellen)
* Agree to wear spectacles for ≥10 hours/day at least 6 days/week.
* Willingness and ability to participate in trial for 3 years and attend scheduled visits.

Exclusion Criteria:

* History of myopia control intervention (e.g., atropine, orthokeratology, multifocal contact lenses, etc.)
* Strabismus by cover test at near or distance wearing correction.
* Amblyopia
* Any ocular or systemic condition known to affect refractive status (e.g., keratoconus, diabetes, Down's syndrome, etc.).
* Current use of ocular or systemic medications which, in the investigator's opinion, may significantly affect pupil size, accommodation or refractive state.
* Current or anticipated use of growth hormones.
* Participation in any clinical study within 30 days of the Baseline visit.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Axial length | 36 Months
  Change in axial length from baseline
Cycloplegic spherical equivalent refraction | 36 Months
  Change in cycloplegic spherical equivalent refraction from baseline

SECONDARY OUTCOMES:
Axial length | 24 Months
  Change in axial length from baseline
Cycloplegic spherical equivalent refraction | 24 Months
  Change in cycloplegic spherical equivalent refraction from baseline

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Scripps Poway Optometry, San Diego, California
  - Sabal Eye Care, Longwood, Florida
  - Illinois College of Optometry, Chicago, Illinois
  - Kannarr Eye Care, Pittsburg, Kansas
  - New England College of Optometry, Boston, Massachusetts
  - SUNY College of Optometry, New York, New York
  - Sacco Eye Group, Vestal, New York
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Mann Eye Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided